CLINICAL TRIAL: NCT05424406
Title: Sleep Reactivity as a Novel Mechanism in Shift Work Disorder
Brief Title: Role of Sleep Reactivity in Shift Work Disorder
Acronym: REACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Philip Cheng, Associate Professor, Henry Ford Health System
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 15661; R01HL160870 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Shift-work Disorder
Keywords: Sleep reactivity
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Two-step mechanistic randomized controlled trial design stratified by high and low sleep reactivity. Step 1: active versus control light therapy; Step 2: Cognitive Behavioral Therapy (CBT) versus sleep education control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active light condition (Experimental): Timed bright light exposure will be delivered in a controlled laboratory setting (10,000 lux) designed to delay the DLMO to 4 am or later. This would shift the circadian nadir (e.g., the period of maximal sleepiness) into the typical daytime sleep period after the nightshift (i.e., circadian nadir at ~10am). Bright light will be delivered in a controlled lab environment using a full spectrum light-box with UV filter (Sunbox Sunray II) to achieve a robust reduction of circadian misalignment. The light schedule will be tailored to each individual nightshift worker, determined by: 1) their baseline circadian phase, and 2) the human phase response curve adjusted to the individual's baseline circadian phase.
  Interventions: Behavioral: Active phototherapy
- Control light condition (Active Comparator): Shift workers randomized to the control condition will receive less intense light that still has a perceptible alerting effect (100 photopic lux). However, light will occur during a portion of the phase response curve with minimal phase shifts.
  Interventions: Behavioral: Control phototherapy
- Cognitive Behavioral Therapy (CBT) condition (Experimental): The CBT condition will probe sleep reactivity using validated CBT strategies over 6 sessions in accordance with the two-factor theory of emotion. Behavioral strategies will be used to reduce physiological arousal (e.g., relaxation training, breathing) and to strengthen behavioral cues for sleep (e.g., sleep hygiene and sleep scheduling). Sleep times will be scheduled to align with the reduced circadian misalignment (compromised phase position, i.e., maintaining a slightly delayed sleep period on offwork days). Cognitive strategies will identify stressors (e.g., dysfunctional beliefs about sleep) and intervene on worry and rumination with cognitive reappraisal and active coping. Sessions will be conducted by a trained behavioral sleep medicine provider via telemedicine to increase accessibility.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Sleep education control condition (Active Comparator): This condition will use an established sleep education control protocol modified for nightshift workers based on the "Plain Language about Shiftwork" published by the National Institute for Occupational Safety and Health (NIOSH). Sleep duration recommendations will be equivalent to the CBT group (8 hours of sleep opportunity) to ensure that outcomes are not confounded by time in bed. Materials in the sleep education control condition will be separated into weekly electronic materials monitored for engagement and completion.
  Interventions: Behavioral: Sleep education control

INTERVENTIONS:
Behavioral: Active phototherapy — Timed bright light exposure delivered in a controlled laboratory setting (10,000 photopic lux) designed to delay the DLMO to 4 am or later.
  Arms: Active light condition
Behavioral: Control phototherapy — Timed less intense light exposure delivered in a controlled laboratory setting (100 photopic lux) that still has a perceptible alerting effect but is not designed to shift circadian phase.
  Arms: Control light condition
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive strategies will identify stressors (e.g., dysfunctional beliefs about sleep) and intervene on worry and rumination with cognitive reappraisal and active coping. Sessions will be conducted by a trained behavioral sleep medicine provider via telemedicine to increase accessibility.
  Arms: Cognitive Behavioral Therapy (CBT) condition
Behavioral: Sleep education control — Sleep duration recommendations will be equivalent to the CBT group (8 hours of sleep opportunity) to ensure that outcomes are not confounded by time in bed. Materials in the sleep education control condition will be separated into weekly electronic materials monitored for engagement and completion.
  Arms: Sleep education control condition

SUMMARY:
The purpose of this project is to test sleep reactivity as an independent cause of Shift Work Disorder (SWD). The primary hypothesis is that those with high sleep reactivity will show persistent SWD symptoms after experimental reduction of circadian misalignment, which will then be mitigated with CBT.

DETAILED DESCRIPTION:
The first aim of this study is to establish sleep reactivity as a predictor of insomnia in SWD independent from circadian misalignment. The second aim of this study is to establish sleep reactivity as a predictor of sleepiness in SWD independent from circadian misalignment. The third aim of this study is to probe sleep reactivity as a cause of insomnia in SWD. The fourth aim of this study is to probe sleep reactivity as a cause of sleepiness in SWD.

Participants with Shift Work Disorder (SWD, N=150) with high and low sleep reactivity will be enrolled. This study will use a two-step mechanistic randomized controlled trial design stratified by high and low sleep reactivity to examine the independent effect of sleep reactivity in SWD after experimental reduction of circadian misalignment. The first step will experimentally reduce circadian misalignment compared to a control. Those who achieve reduced circadian misalignment (melatonin onset at or later than 4am, i.e., compromised phase position) and remain symptomatic will continue to the second step where sleep reactivity will be probed with CBT compared to a sleep education control.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be working a fixed nightshift schedule, operationalized as: a) working at least three night shifts a week, b) shifts must begin between 18:00 and 02:00, and last between 8 to 12 hours, and c) must also plan to maintain the nightshift schedule for the duration of the study
* Participants must have Shift Work Disorder, which will be diagnosed based on ICSD-3 criteria
* Participants must show circadian misalignment, operationalized as a baseline melatonin onset between 18:00 and 01:00.
* Participants must be at least 18 years old

Exclusion Criteria:

* Insomnia disorder or excessive sleepiness predating the onset of shift work
* Termination of nightshift schedule
* Presence of other sleep disorders (e.g. obstructive sleep apnea, narcolepsy) determined by standard clinical polysomnography
* Diagnosis of bipolar disorder
* History of neurological disorders determined by self-report and medical history
* Pregnancy
* Alcohol use disorder
* Illicit drug use via self-report and urine drug screen if reasonable suspicion to test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Dim light melatonin onset | Within two days of treatment for a duration of 24 hours
  Melatonin values will be measured in saliva samples, collected in dim light conditions in a laboratory, to determine circadian phase.
Sleep reactivity | Within two weeks of treatment
  Sleep reactivity will be measured using the validated Ford Insomnia Response to Stress Test (FIRST). Based on psychometric testing of the FIRST, a cutoff score of 16 will distinguish high and low sleep reactivity.

SECONDARY OUTCOMES:
Insomnia | Within one week of post-treatment
  Insomnia will be measured with the Insomnia Severity Scale (0 to 28; higher scores correspond to worse severity)
Sleepiness | Within one week of post-treamtnet
  Sleepiness will be measured with the Epworth Sleepiness Scale (0 to 24; a score of 10 or greater indicates excessive sleepiness).

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Columbus Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Request for data sharing will be evaluated on a case-by-case basis.